CLINICAL TRIAL: NCT02352116
Title: Evaluation of Post-PACU Pain Management Experiences in Pediatric Ambulatory Surgery Patients
Brief Title: Evaluation of Post-PACU Pain Management in Pediatric Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Lena S. Sun, Emanuel M. Papper Professor of Anesthesiology and Professor of Pediatrics, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: AAAI5954
Record Dates: First submitted 2014-11-21; First posted 2015-02-02 (Estimated); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Pain
Keywords: Postoperative Experience; Postoperative Behavioral Changes; Maladaptive Behavioral Changes
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Additional education (Experimental): Subjects undergoing ambulatory surgery who receive standard of care management with additional face-to-face education in postoperative pain management.
  Interventions: Other: Additional face-to-face education; Other: Standard of care management
- No additional education (Active Comparator): Subjects undergoing ambulatory surgery who receive standard of care management with no additional education in postoperative pain management.
  Interventions: Other: Standard of care management

INTERVENTIONS:
Other: Additional face-to-face education — Additional teaching regarding what to expect in terms of postoperative pain, how to properly identify pain in children, and instruction on the proper administration of analgesic medications
  Arms: Additional education
Other: Standard of care management — Current standard of care at a major U.S. teaching hospital.

SUMMARY:
This study aims to assess the differences in overall pain severity, pain management, and satisfaction during recovery period between two groups of children who either receive or do not receive additional education related to expectation and management of postoperative pain.

DETAILED DESCRIPTION:
With the increased frequency and popularity of pediatric ambulatory surgery, there is a greater need for evaluation of the postoperative pain experience after discharge from the hospital. Pain is one of the most significant factors affecting the postoperative experience in adults, and also be true in the pediatric population. Control of postoperative pain in children after discharge from the hospital poses particular challenges due to dependence on parental or caretaker ability to properly evaluate the child's pain, their understanding of appropriate dosing of pain medications, and their willingness to administer enough medications until sufficient relief is achieved.

The investigators aim to assess the differences in reported pain between groups who receive additional face-to-face education versus the current standard of care at a major US teaching hospital. The study will assess pain management after surgery using parental reports and questionnaires to assess their child's pain at multiple time points during the study. Additionally, this study will also assess baseline behavioral attributes of children and will compare behavioral changes at 24-48 hours, 7-10 days, and 2-4 weeks postoperatively as these behavior changes may also affect overall postoperative experience.

This study is divided into phase I and phase II. Phase I is the initial assessment of the investigators' institution's pain management in healthy pediatric patients undergoing ambulatory surgical procedures. Phase II consists of randomized trial which includes a randomized intervention group and control group. The group selected randomly for intervention will receive additional teaching regarding what to expect in terms of postoperative pain and how to properly identify pain in children.

ELIGIBILITY:
Inclusion Criteria:

* Patients ages 1-6 years undergoing ambulatory surgical procedures.
* Patients with an ASA status of I or II spending 23 hours or less recovering in the PACU and discharged home.

Exclusion Criteria:

* Patients with an ASA status of III or IV.
* Patients admitted as inpatients or transferred to the PICU or inpatient for recovery, and any conditions that may affect pain expression or sensation.

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 900 (Estimated)
Dates: Start 2013-06 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Postoperative Pain Measure for Parents Score | baseline, 72 hours, 7-14 days, up to 4 weeks
  Validated questionnaire for parental assessment of pain in children ages 1-12 years

SECONDARY OUTCOMES:
Change in Postoperative Anesthesia Emergence Delirium (PAED) Score | baseline, 72 hours, 7-14 days, up to 4 weeks
  Validated 5-question survey completed by nurses after arrival in the post-operative anesthesia unit
Change in Emotionality, Activity, Sociability, Impulsivity Instrument of child Temperament (EASI) Scale | baseline, 72 hours, 7-14 days, up to 4 weeks
  The EASI is a parent report form that assesses a child's baseline temperament and yields subscales including emotionality and activity level.
  The scale contains 14 items to which participants respond on a 5- point Likert scale ranging from "Strongly disagree" to "Strongly agree". Higher scores indicate greater emotionality.
Change in Modified Yale Preoperative Anxiety Scale (mYPAS) | baseline, 72 hours, 7-14 days, up to 4 weeks
  An observational measure of children's preoperative anxiety. Contains 27 items that measure activity, emotional expressivity, state of arousal, vocalization, use of parents. This must be administered by trained research assistants. Validated for children ages 2 and older
Change in Post-Hospital Behavior Questionnaire Score | baseline, 72 hours, 7-14 days, up to 4 weeks
  A validated questionnaire to be completed by the parents. This measure contains 27 items that evaluate a child's general anxiety, separation anxiety, anxiety about sleep, easting disturbance, aggression toward authority, and apathy/withdrawal

CONTACTS AND LOCATIONS:
Overall Officials: Lena S. Sun, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States